CLINICAL TRIAL: NCT00203021
Title: Open Label Study to Evaluate the Safety of Copaxone® and to Monitor the Neurologic Course of Disease in Multiple Sclerosis Patients Treated With Copaxone
Brief Title: Glatiramer Acetate (Copaxone®) Study to Follow Participants From the First Original Study for Safety and Effectiveness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GA-9004; 01-9004 (Other: Teva)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2019-07-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Glatiramer Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Glatiramer Acetate: Delayed Start (Experimental): Participants who were originally randomized to the placebo group in the 01-9001 and/or the 01-9001E studies received glatiramer acetate 20 milligrams (mg) subcutaneous (SC) injection daily at the start of this study. After 18 July 2014 (protocol amendment 12), participants were offered the opportunity to continue treatment with glatiramer acetate 20 mg daily or switch to glatiramer acetate 40 mg three times weekly (TIW). The treatment continued for up to 288 months.
  Interventions: Drug: Glatiramer acetate
- Glatiramer Acetate: Early Start (Experimental): Participants who were originally randomized to the glatiramer acetate 20 mg group in the 01-9001 and/or the 01-9001E studies continued to receive glatiramer acetate 20 mg SC injection daily at the start of this study. After 18 July 2014 (protocol amendment 12), participants were offered the opportunity to continue treatment with glatiramer acetate 20 mg daily or switch to glatiramer acetate 40 mg TIW. The treatment continued for up to 288 months.
  Interventions: Drug: Glatiramer acetate

INTERVENTIONS:
Drug: Glatiramer acetate — Glatiramer acetate will be administered as per the dose and schedule specified in the respective arms.
  Other Names: Copaxone®

SUMMARY:
This open-label extension study will evaluate the long-term safety of glatiramer acetate and its effect on the neurologic course of participants with relapsing-remitting multiple sclerosis (RRMS). Participants have scheduled visits every 3 months to assess glatiramer acetate safety and their Multiple Sclerosis (MS) status.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have participated (been randomized) in the Copaxone double-blind placebo-controlled study 01-9001 and/or the double-placebo-controlled extension study 01-9001E.
* Participants could be male or female. Women of childbearing potential must have practiced an acceptable method of birth control.
* Participants must have completed the scheduled termination visit for Amendment 12 (Month 264).
* Participants must have signed an approved informed consent form (ICF) prior to continuing in the study extension or at the first visit in the extension (Month 264 which corresponds to the termination visit of Amendment 12).
* Participants must have been psychologically and physically stable to participate in the trial as judged by the investigator.
* All participants enrolled in this extension study were required to have the following study-specific baseline characteristics prior to entry to Study 01-9001: a diagnosis of RRMS as defined by Poser et al 1983, at least 2 clearly identified relapses and remissions in the 2-year period prior to study entry, ambulatory with a Kurtzke EDSS score of 0 to 5.0 inclusive, and a stable neurologic state for at least 30 days prior to study entry.

Exclusion Criteria:

* Pregnancy or lactation.
* Medical or psychiatric conditions that affect the participant's ability to give informed consent or complete the study.
* Inability to self-administer subcutaneous medication or lack of another responsible individual to administer the study preparation daily.
* Use of approved MS therapies including interferons, experimental MS therapies, or previous immunosuppressive therapy with cytotoxic chemotherapy (azathioprine, cyclophosphamide, or cyclosporine).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 1994-03-26 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cory Ford, MD, Study Director — University of New Mexico
Locations (11):
- United States (11):
  - Teva Investigational Site 009, Los Angeles, California
  - Teva Investigational Site 004, Los Angeles, California
  - Teva Investigational Site 008, New Haven, Connecticut
  - Teva Investigational Site 005, Baltimore, Maryland
  - Teva Investigational Site 003, Detroit, Michigan
  - Teva Investigational Site 002, Albuquerque, New Mexico
  - Teva Investigational Site 007, Rochester, New York
  - Teva Investigational Site 001, Philadelphia, Pennsylvania
  - Teva Investigational Site 010, Houston, Texas
  - Teva Investigational Site 006, Salt Lake City, Utah
  - Teva Investigational Site 011, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who participated in both or either Studies 01-9001 (double-blind [DB] placebo-controlled study) and 01-9001E (DB extension study) were eligible to enter into this open-label extension study. Note that the 01-9001 and 01-9001E studies predate NCT assignments.
Pre-assignment Details: A total of 209 participants were screened; 208 participants met entry criteria and were enrolled in this study.
Period: Overall Study
Arm/Group | Glatiramer Acetate: Delayed Start | Glatiramer Acetate: Early Start
Started | 107 | 101
Received at Least 1 Dose of Study Drug | 107 | 101
Completed | 28 | 24
Not Completed | 79 | 77
Not completed — Death | 4 | 1
Not completed — Adverse Event | 10 | 5
Not completed — Withdrawal by Subject | 45 | 48
Not completed — Lost to Follow-up | 9 | 7
Not completed — Other than specified | 11 | 16

BASELINE CHARACTERISTICS:
Population: 01-9004 included participants originally randomized to placebo in 01-9001 and/or 01-9001E studies and switched to glatiramer acetate 20 mg at the start of the 01-9004 study; and participants originally randomized to the glatiramer acetate 20 mg group in 01-9001 and/or 01-9001E studies who continued on this dose in the 01-9004 study.
Groups:
- Glatiramer Acetate: Delayed Start: Participants who were originally randomized to the placebo group in the 01-9001 and/or the 01-9001E studies received glatiramer acetate 20 mg SC injection daily at the start of this study. After 18 July 2014 (protocol amendment 12), participants were offered the opportunity to continue treatment with glatiramer acetate 20 mg daily or switch to glatiramer acetate 40 mg TIW. The treatment continued for up to 288 months.
- Total: Total of all reporting groups
Arm/Group | Glatiramer Acetate: Delayed Start | Glatiramer Acetate: Early Start | Total
Number analyzed (Participants) | 107 | 101 | 208
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.9 (6.57) | 37.2 (5.79) | 37.1 (6.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 72 | 154
  Male | 25 | 29 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 105 | 101 | 206
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 101 | 97 | 198
  Black | 2 | 3 | 5
  American Indian or Alaskan Native | 1 | 1 | 2
  Other | 1 | 0 | 1
  Missing | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious AEs were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. Any AEs included both serious and non-serious AEs. A summary of other non-serious AEs and all serious AEs, regardless of causality, is located in Reported AE section.
Time Frame: Baseline up to Month 288
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Glatiramer Acetate: Delayed Start | Glatiramer Acetate: Early Start
Number analyzed (Participants) | 107 | 101
participants
  Any AEs | 107 | 100
  Serious AEs | 44 | 38

2. Primary Outcome: Change From Baseline in Kurtzke Expanded Disability Status Scale (EDSS) Score at Month 288
Description: The EDSS uses an ordinal scale to assess neurologic impairment in Multiple Sclerosis based on a neurological examination. Scores in each of 7 functional systems (Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel and Bladder, and Cerebral) and an ambulation score were combined to determine the total EDSS score, ranging from 0 (normal) to 10 (death due to Multiple Sclerosis).
Time Frame: Baseline, Month 288
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Glatiramer Acetate: Delayed Start | Glatiramer Acetate: Early Start
Number analyzed (Participants) | 28 | 24
units on a scale
  Baseline | 2.34 (1.599) | 2.23 (1.406)
  Change at Month 288 | 1.64 (1.962) | 1.06 (1.896)

ADVERSE EVENTS:
Time Frame: Baseline up to Month 288
Description: 01-9004 included participants originally randomized to placebo in 01-9001 and/or 01-9001E studies and switched to glatiramer acetate 20 mg at the start of the 01-9004 study; and participants originally randomized to the glatiramer acetate 20 mg group in 01-9001 and/or 01-9001E studies who continued on this dose in the 01-9004 study.
Arm/Group | Glatiramer Acetate: Delayed Start | Glatiramer Acetate: Early Start
All-Cause Mortality (participants affected / at risk) | 4/107 | 1/101
Serious Adverse Events (participants affected / at risk) | 44/107 | 38/101
Other Adverse Events (participants affected / at risk) | 107/107 | 100/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glatiramer Acetate: Delayed Start (N=107) | Glatiramer Acetate: Early Start (N=101)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 3 (3)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (3) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (2)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Diverticulitis Meckel's (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Thyroid cyst (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Adhesion (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (3) | 5 (6)
Complication associated with device (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Facial pain (General disorders) | 1 (1) | 0 (0)
Feeling abnormal (General disorders) | 1 (1) | 0 (0)
Haemorrhagic cyst (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Injection site inflammation (General disorders) | 1 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Strangulated hernia (General disorders) | 1 (1) | 0 (0)
Biliary cirrhosis primary (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (5)
Catheter site abscess (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Kidney infection (Infections and infestations) | 0 (0) | 2 (2)
Mastitis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis aseptic (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Post procedural sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 2 (3) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (7) | 4 (4)
Wound infection fungal (Infections and infestations) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Failure to anastomose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (3) | 1 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Cardiac output decreased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 5 (6) | 2 (3)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung carcinoma cell type unspecified stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (5)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Drug withdrawal convulsions (Nervous system disorders) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 1 (1) | 1 (1)
Multiple sclerosis relapse (Nervous system disorders) | 1 (1) | 0 (0)
Muscle spasticity (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 2 (2)
Seizure (Nervous system disorders) | 3 (3) | 0 (0)
Sensory loss (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient global amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 2 (2) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Anger (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 5 (8)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Calculus urethral (Renal and urinary disorders) | 1 (1) | 0 (0)
Neurogenic bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Breast disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 2 (3) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Pelvic adhesions (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Rectocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Appendicectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Bladder repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Central venous catheterisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Femoral hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 2 (2) | 2 (2)
Hysterosalpingo-oophorectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Small intestinal resection (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal laminectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (2)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glatiramer Acetate: Delayed Start (N=107) | Glatiramer Acetate: Early Start (N=101)
Anaemia (Blood and lymphatic system disorders) | 11 (11) | 9 (9)
Lymphadenopathy (Blood and lymphatic system disorders) | 10 (23) | 7 (57)
Palpitations (Cardiac disorders) | 12 (31) | 9 (28)
Tachycardia (Cardiac disorders) | 6 (13) | 8 (21)
Ear pain (Ear and labyrinth disorders) | 7 (10) | 11 (14)
Tinnitus (Ear and labyrinth disorders) | 11 (16) | 10 (14)
Vertigo (Ear and labyrinth disorders) | 18 (28) | 16 (31)
Hypothyroidism (Endocrine disorders) | 4 (4) | 6 (7)
Diplopia (Eye disorders) | 14 (18) | 9 (12)
Dry eye (Eye disorders) | 6 (8) | 2 (3)
Eye pain (Eye disorders) | 6 (11) | 16 (32)
Vision blurred (Eye disorders) | 24 (37) | 19 (33)
Visual acuity reduced (Eye disorders) | 4 (5) | 9 (12)
Visual impairment (Eye disorders) | 13 (16) | 9 (11)
Abdominal discomfort (Gastrointestinal disorders) | 13 (19) | 13 (16)
Abdominal pain (Gastrointestinal disorders) | 10 (21) | 16 (25)
Abdominal pain upper (Gastrointestinal disorders) | 8 (11) | 6 (6)
Anal incontinence (Gastrointestinal disorders) | 11 (18) | 12 (28)
Constipation (Gastrointestinal disorders) | 23 (38) | 20 (30)
Defaecation urgency (Gastrointestinal disorders) | 5 (11) | 6 (8)
Diarrhoea (Gastrointestinal disorders) | 25 (45) | 27 (48)
Dyspepsia (Gastrointestinal disorders) | 12 (22) | 10 (14)
Dysphagia (Gastrointestinal disorders) | 11 (17) | 8 (16)
Gastritis (Gastrointestinal disorders) | 6 (9) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 12 (15) | 14 (16)
Hiatus hernia (Gastrointestinal disorders) | 1 (4) | 6 (7)
Large intestine polyp (Gastrointestinal disorders) | 6 (6) | 5 (5)
Nausea (Gastrointestinal disorders) | 31 (66) | 24 (59)
Toothache (Gastrointestinal disorders) | 6 (8) | 6 (9)
Vomiting (Gastrointestinal disorders) | 16 (22) | 14 (28)
Asthenia (General disorders) | 8 (9) | 13 (19)
Chest discomfort (General disorders) | 17 (64) | 13 (66)
Chest pain (General disorders) | 12 (15) | 6 (9)
Chills (General disorders) | 9 (26) | 5 (6)
Fatigue (General disorders) | 58 (145) | 59 (159)
Feeling hot (General disorders) | 5 (6) | 6 (11)
Gait disturbance (General disorders) | 14 (20) | 18 (25)
Ill-defined disorder (General disorders) | 8 (9) | 3 (4)
Injection site bruising (General disorders) | 11 (18) | 6 (9)
Injection site erythema (General disorders) | 68 (87) | 33 (40)
Injection site haemorrhage (General disorders) | 8 (12) | 4 (5)
Injection site induration (General disorders) | 20 (28) | 6 (18)
Injection site mass (General disorders) | 26 (68) | 14 (24)
Injection site pain (General disorders) | 52 (111) | 15 (19)
Injection site pruritus (General disorders) | 25 (29) | 11 (15)
Injection site reaction (General disorders) | 8 (11) | 4 (5)
Injection site swelling (General disorders) | 34 (43) | 11 (12)
Injection site urticaria (General disorders) | 12 (28) | 8 (8)
Injection site warmth (General disorders) | 10 (14) | 4 (4)
Oedema peripheral (General disorders) | 10 (13) | 7 (10)
Pain (General disorders) | 16 (31) | 8 (12)
Peripheral swelling (General disorders) | 13 (16) | 8 (10)
Pyrexia (General disorders) | 11 (23) | 15 (21)
Hypersensitivity (Immune system disorders) | 8 (9) | 8 (11)
Seasonal allergy (Immune system disorders) | 15 (24) | 13 (22)
Bronchitis (Infections and infestations) | 20 (35) | 22 (44)
Cellulitis (Infections and infestations) | 7 (9) | 6 (7)
Conjunctivitis (Infections and infestations) | 8 (13) | 5 (5)
Cystitis (Infections and infestations) | 13 (24) | 5 (5)
Ear infection (Infections and infestations) | 11 (13) | 9 (12)
Fungal infection (Infections and infestations) | 9 (11) | 13 (27)
Gastroenteritis (Infections and infestations) | 7 (7) | 5 (7)
Gastroenteritis viral (Infections and infestations) | 17 (22) | 16 (24)
Herpes zoster (Infections and infestations) | 7 (12) | 10 (12)
Influenza (Infections and infestations) | 33 (55) | 25 (40)
Nasopharyngitis (Infections and infestations) | 32 (98) | 28 (74)
Oral herpes (Infections and infestations) | 7 (12) | 6 (15)
Pharyngitis (Infections and infestations) | 6 (9) | 4 (4)
Pharyngitis streptococcal (Infections and infestations) | 9 (9) | 7 (7)
Pneumonia (Infections and infestations) | 9 (10) | 9 (11)
Sinusitis (Infections and infestations) | 37 (115) | 37 (108)
Tooth abscess (Infections and infestations) | 10 (10) | 5 (7)
Tooth infection (Infections and infestations) | 3 (5) | 9 (10)
Upper respiratory tract infection (Infections and infestations) | 66 (283) | 64 (282)
Urinary tract infection (Infections and infestations) | 51 (281) | 48 (248)
Vaginal infection (Infections and infestations) | 5 (13) | 7 (7)
Vulvovaginal mycotic infection (Infections and infestations) | 9 (19) | 11 (18)
Contusion (Injury, poisoning and procedural complications) | 27 (49) | 20 (28)
Fall (Injury, poisoning and procedural complications) | 31 (78) | 35 (79)
Foot fracture (Injury, poisoning and procedural complications) | 15 (21) | 13 (15)
Hand fracture (Injury, poisoning and procedural complications) | 9 (9) | 6 (7)
Joint injury (Injury, poisoning and procedural complications) | 3 (3) | 9 (10)
Laceration (Injury, poisoning and procedural complications) | 13 (17) | 13 (16)
Ligament sprain (Injury, poisoning and procedural complications) | 11 (13) | 12 (15)
Muscle strain (Injury, poisoning and procedural complications) | 9 (11) | 13 (13)
Post procedural complication (Injury, poisoning and procedural complications) | 8 (12) | 3 (8)
Procedural pain (Injury, poisoning and procedural complications) | 14 (31) | 13 (24)
Rib fracture (Injury, poisoning and procedural complications) | 4 (4) | 7 (8)
Road traffic accident (Injury, poisoning and procedural complications) | 6 (8) | 6 (6)
Skin abrasion (Injury, poisoning and procedural complications) | 8 (15) | 7 (8)
Weight decreased (Investigations) | 7 (15) | 4 (6)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 9 (13) | 14 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 32 (60) | 34 (91)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (5) | 7 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 34 (82) | 36 (74)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (8) | 6 (8)
Joint swelling (Musculoskeletal and connective tissue disorders) | 7 (11) | 6 (9)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 4 (4) | 10 (16)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 20 (35) | 24 (47)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 7 (12) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 45 (81) | 38 (78)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 18 (27) | 12 (16)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 17 (35) | 19 (34)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 9 (15)
Neck pain (Musculoskeletal and connective tissue disorders) | 17 (25) | 8 (13)
Osteopenia (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (7)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 9 (12) | 9 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 33 (72) | 37 (73)
Tendonitis (Musculoskeletal and connective tissue disorders) | 6 (9) | 5 (11)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (7) | 4 (4)
Amnesia (Nervous system disorders) | 5 (10) | 8 (14)
Balance disorder (Nervous system disorders) | 23 (50) | 27 (47)
Burning sensation (Nervous system disorders) | 9 (17) | 10 (28)
Cognitive disorder (Nervous system disorders) | 8 (11) | 6 (8)
Coordination abnormal (Nervous system disorders) | 5 (6) | 7 (11)
Dizziness (Nervous system disorders) | 39 (85) | 29 (56)
Dysaesthesia (Nervous system disorders) | 7 (8) | 7 (10)
Dysarthria (Nervous system disorders) | 10 (19) | 9 (12)
Headache (Nervous system disorders) | 46 (89) | 40 (96)
Hemiparesis (Nervous system disorders) | 6 (7) | 8 (10)
Hyperaesthesia (Nervous system disorders) | 6 (19) | 6 (6)
Hypoaesthesia (Nervous system disorders) | 41 (97) | 42 (106)
Memory impairment (Nervous system disorders) | 12 (20) | 9 (15)
Migraine (Nervous system disorders) | 9 (14) | 13 (25)
Muscle spasticity (Nervous system disorders) | 16 (21) | 23 (38)
Optic neuritis (Nervous system disorders) | 6 (6) | 5 (8)
Paraesthesia (Nervous system disorders) | 33 (66) | 32 (75)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 7 (10)
Sensory disturbance (Nervous system disorders) | 6 (9) | 5 (8)
Sinus headache (Nervous system disorders) | 4 (5) | 7 (7)
Tremor (Nervous system disorders) | 16 (39) | 9 (33)
Visual field defect (Nervous system disorders) | 2 (2) | 6 (6)
Affect lability (Psychiatric disorders) | 6 (16) | 6 (10)
Anxiety (Psychiatric disorders) | 30 (53) | 28 (65)
Depression (Psychiatric disorders) | 33 (86) | 40 (118)
Emotional distress (Psychiatric disorders) | 4 (13) | 8 (21)
Insomnia (Psychiatric disorders) | 33 (90) | 36 (92)
Stress (Psychiatric disorders) | 4 (5) | 6 (10)
Dysuria (Renal and urinary disorders) | 9 (13) | 7 (14)
Micturition urgency (Renal and urinary disorders) | 22 (41) | 31 (60)
Pollakiuria (Renal and urinary disorders) | 18 (35) | 26 (35)
Urinary hesitation (Renal and urinary disorders) | 8 (9) | 10 (15)
Urinary incontinence (Renal and urinary disorders) | 17 (38) | 12 (28)
Urinary retention (Renal and urinary disorders) | 7 (17) | 11 (16)
Erectile dysfunction (Reproductive system and breast disorders) | 4 (4) | 6 (16)
Menorrhagia (Reproductive system and breast disorders) | 6 (9) | 5 (5)
Menstruation irregular (Reproductive system and breast disorders) | 10 (30) | 7 (12)
Metrorrhagia (Reproductive system and breast disorders) | 6 (9) | 2 (4)
Vaginal haemorrhage (Reproductive system and breast disorders) | 4 (6) | 6 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (25) | 12 (22)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 (68) | 11 (25)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 9 (21)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 22 (41) | 14 (26)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 4 (6)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (7)
Acne (Skin and subcutaneous tissue disorders) | 6 (9) | 7 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (13) | 4 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (10) | 1 (2)
Erythema (Skin and subcutaneous tissue disorders) | 16 (18) | 9 (12)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6 (7) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (11) | 6 (14)
Rash (Skin and subcutaneous tissue disorders) | 17 (26) | 21 (34)
Urticaria (Skin and subcutaneous tissue disorders) | 7 (8) | 8 (14)
Tooth extraction (Surgical and medical procedures) | 7 (9) | 1 (1)
Flushing (Vascular disorders) | 22 (104) | 9 (67)
Hot flush (Vascular disorders) | 4 (7) | 6 (12)
Hypertension (Vascular disorders) | 11 (14) | 15 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-13): https://cdn.clinicaltrials.gov/large-docs/21/NCT00203021/Prot_SAP_000.pdf